CLINICAL TRIAL: NCT03314519
Title: A Randomized Controlled Study Compare Lung Ultrasonography to Fiberoptic Bronchoscopy Confirming Double Lumen Tube Positioning for Thoracic Surgery.
Brief Title: Lung Ultrasonography vs Fiberoptic Bronchoscopy for Aiding Lung Collapse in Patient Using Double Lumen Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Skanavitoon
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Lung Diseases; Ultrasonography; Fiberoptic Bronchoscopy; One Lung Ventilation; Thoracic Surgery; Lung Collapse
Keywords: Lung ultrasonography; Lung collapse; fiberoptic bronchoscopy; double lumen tube; compare; one lung ventilation; thoracic surgery; thoracic anaesthesia; lung ultrasound
MeSH Terms: conditions — Lung Diseases; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Compare lung collapse of lung ultrasonography to fiberoptic bronchoscopy.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultrasonography (Experimental): Patients in this group receive lung ultrasonography to detect lung collapse after insert double lumen tube and finally compare lung collapse by the surgeon's visual grading scale of lung collapse when entering pleural cavity.
  Interventions: Diagnostic Test: Lung ultrasonography by experienced anaesthesiologist
- Fiberoptic bronchoscopy (Active Comparator): Patients in this group receive fiberoptic bronchoscope to detect lung collapse after inserting a double lumen tube and finally compare lung collapse by the surgeon's visual grading scale of lung collapse when entering the pleural cavity.
  Interventions: Diagnostic Test: Fiberoptic bronchoscopy for double lumen tube's position

INTERVENTIONS:
Diagnostic Test: Lung ultrasonography by experienced anaesthesiologist — Use ultrasound image of lung at upper and lower lobe to detect lung collapse and compare grading of lung collapse by surgeon as gold standard
  Arms: Ultrasonography
Diagnostic Test: Fiberoptic bronchoscopy for double lumen tube's position — Use fiberoptic bronchoscope via double lumen tube to detect optimum position of double lumen tube and record grading of lung collapse by surgeon as gold standard
  Arms: Fiberoptic bronchoscopy

SUMMARY:
The study contains the result from a comparison of diagnostic outcomes about lung collapse by using lung ultrasonography as a new diagnostic test compares to fiberoptic bronchoscopy as the standard test.

DETAILED DESCRIPTION:
The study contains the result from a comparison of diagnostic outcomes about lung collapse by using lung ultrasonography as a new diagnostic test compares to fiberoptic bronchoscopy as a standard test. Both of them detect lung collapse reported as surgical grading lung collapse by the thoracic surgeons. The protocol was performed in a randomized controlled trial whether the subject was allocated to the ultrasonography group or the fiberoptic bronchoscopy group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥18 years old
* American Society of Anesthesiologists(ASA) physical status classification I - III
* Scheduled for elective thoracic surgery which requires One lung ventilation(OLV) with Left-sided double lumen tube

Exclusion Criteria:

* Anticipated difficult intubation or with the tracheostomy tube
* Patient with pneumothorax, pleural effusion, emphysema or past history of pleurodesis
* Patient with deranges pulmonary function test (out of forced expiration volume in 1 s, total lung capacity, forced vital capacity <50% of the predicted values)
* The patient refuses to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kasana Raksamani, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bussieres JS, Somma J, Del Castillo JL, Lemieux J, Conti M, Ugalde PA, Gagne N, Lacasse Y. Bronchial blocker versus left double-lumen endotracheal tube in video-assisted thoracoscopic surgery: a randomized-controlled trial examining time and quality of lung deflation. Can J Anaesth. 2016 Jul;63(7):818-27. doi: 10.1007/s12630-016-0657-3. Epub 2016 May 2. PMID 27138896
- [Background] Boucek CD, Landreneau R, Freeman JA, Strollo D, Bircher NG. A comparison of techniques for placement of double-lumen endobronchial tubes. J Clin Anesth. 1998 Nov;10(7):557-60. doi: 10.1016/s0952-8180(98)00081-6. PMID 9805696
- [Background] Alvarez-Diaz N, Amador-Garcia I, Fuentes-Hernandez M, Dorta-Guerra R. Comparison between transthoracic lung ultrasound and a clinical method in confirming the position of double-lumen tube in thoracic anaesthesia. A pilot study. Rev Esp Anestesiol Reanim. 2015 Jun-Jul;62(6):305-12. doi: 10.1016/j.redar.2014.06.005. Epub 2014 Aug 20. English, Spanish. PMID 25149114
- [Background] Cohen E. Double-lumen tube position should be confirmed by fiberoptic bronchoscopy. Curr Opin Anaesthesiol. 2004 Feb;17(1):1-6. doi: 10.1097/00001503-200402000-00002. PMID 17021522
- [Background] Parab SY, Divatia JV, Chogle A. A prospective comparative study to evaluate the utility of lung ultrasonography to improve the accuracy of traditional clinical methods to confirm position of left sided double lumen tube in elective thoracic surgeries. Indian J Anaesth. 2015 Aug;59(8):476-81. doi: 10.4103/0019-5049.162983. PMID 26379290
- [Background] Diaz NG. "A prospective comparative study to evaluate the utility of lung ultrasonography to improve the accuracy of traditional clinical methods to confirm position of left sided double lumen tube in elective thoracic surgeries". Indian J Anaesth. 2016 Mar;60(3):226-7. doi: 10.4103/0019-5049.177880. No abstract available. PMID 27053795
- [Background] Lohser J. Evidence-based management of one-lung ventilation. Anesthesiol Clin. 2008 Jun;26(2):241-72, v. doi: 10.1016/j.anclin.2008.01.011. PMID 18456211
- [Background] Kitabjian L, Bordi S, Elisha S, Gabot M, Heiner J, Nagelhout J, Thompson J. Anesthesia case management for video-assisted thoracoscopic surgery. AANA J. 2013 Feb;81(1):65-72. PMID 23513327
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376
- [Background] Yamaguchi Y, Moharir A, Burrier C, Tobias JD. Point-of-care lung ultrasound to evaluate lung isolation during one-lung ventilation in children: A case report. Saudi J Anaesth. 2019 Jul-Sep;13(3):243-245. doi: 10.4103/sja.SJA_115_19. PMID 31333372
- [Background] Nam JS, Park I, Seo H, Min HG. The use of lung ultrasonography to confirm lung isolation in an infant who underwent emergent video-assisted thoracoscopic surgery: a case report. Korean J Anesthesiol. 2015 Aug;68(4):411-4. doi: 10.4097/kjae.2015.68.4.411. Epub 2015 Jul 28. PMID 26257857
- [Background] Saporito A, Lo Piccolo A, Franceschini D, Tomasetti R, Anselmi L. Thoracic ultrasound confirmation of correct lung exclusion before one-lung ventilation during thoracic surgery. J Ultrasound. 2013 Nov 9;16(4):195-9. doi: 10.1007/s40477-013-0050-9. eCollection 2013 Nov 9. PMID 24432174
- [Background] See KC, Ong V, Wong SH, Leanda R, Santos J, Taculod J, Phua J, Teoh CM. Lung ultrasound training: curriculum implementation and learning trajectory among respiratory therapists. Intensive Care Med. 2016 Jan;42(1):63-71. doi: 10.1007/s00134-015-4102-9. Epub 2015 Oct 16. PMID 26474994
- [Background] de Bellis M, Accardo R, Di Maio M, La Manna C, Rossi GB, Pace MC, Romano V, Rocco G. Is flexible bronchoscopy necessary to confirm the position of double-lumen tubes before thoracic surgery? Eur J Cardiothorac Surg. 2011 Oct;40(4):912-6. doi: 10.1016/j.ejcts.2011.01.070. Epub 2011 Jul 29. PMID 21802958
- [Background] Chou EH, Dickman E, Tsou PY, Tessaro M, Tsai YM, Ma MH, Lee CC, Marshall J. Ultrasonography for confirmation of endotracheal tube placement: a systematic review and meta-analysis. Resuscitation. 2015 May;90:97-103. doi: 10.1016/j.resuscitation.2015.02.013. Epub 2015 Feb 21. PMID 25711517
- [Background] Sustic A, Protic A, Cicvaric T, Zupan Z. The addition of a brief ultrasound examination to clinical assessment increases the ability to confirm placement of double-lumen endotracheal tubes. J Clin Anesth. 2010 Jun;22(4):246-9. doi: 10.1016/j.jclinane.2009.07.010. PMID 20522353
- [Background] Parab SY, Kumar P, Divatia JV, Sharma K. A prospective randomized controlled double-blind study comparing auscultation and lung ultrasonography in the assessment of double lumen tube position in elective thoracic surgeries involving one lung ventilation at a tertiary care cancer institute. Korean J Anesthesiol. 2019 Feb;72(1):24-31. doi: 10.4097/kja.d.17.00081. Epub 2018 Sep 12. PMID 30205667
- [Derived] Kanavitoon S, Raksamani K, Troy MP, Suphathamwit A, Thongcharoen P, Suksompong S, Oh SS. Lung ultrasound is non-inferior to bronchoscopy for confirmation of double-lumen endotracheal tube positioning: a randomized controlled noninferiority study. BMC Anesthesiol. 2022 May 30;22(1):168. doi: 10.1186/s12871-022-01707-4. PMID 35637457

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy
Started | 100 | 100
Completed | 97 | 98
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Population: There are protocol deviations of 3 patients in Group US and 2 patients in group FOB.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There are protocol deviations of 3 patients in Group US and 2 patients in group FOB.
  years | 60.4 (15.6) | 60.6 (12.8) | 60.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are protocol deviations of 3 patients in Group US and 2 patients in group FOB.
  Participants
    Female | 59 | 50 | 109
    Male | 38 | 48 | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Thailand | 97 | 98 | 195
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (4.4) | 24.0 (4.3) | 24.2 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients of Lung Collapse in Ultrasonography and Fiberoptic Bronchoscopy
Description: Compare number of patients with lung collapse detected by ultrasonography and fiberoptic bronchoscopy in patient with double lumen tube by report as specificity and sensitivity of detection of lung collapse by compare to visual grading of lung collapse by surgeon
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy
Number analyzed (Participants) | 97 | 98
Participants | 89 | 83

2. Secondary Outcome: Timing to Detect Lung Collapse
Description: Time point from evaluation of lung collapse by each test to time point of grading lung collapse by gold standard( visual grading of lung collapse by surgeon)
Time Frame: 30 minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy
Number analyzed (Participants) | 97 | 98
minutes | 14 [9.5 to 20] | 9 [5 to 14.3]

3. Secondary Outcome: Accuracy of Detection of Lung Collapse in Ultrasonography Method in Cardiovascular and Thoracic Anesthesia Fellow
Description: Accuracy of detection of lung collapse in thoracic patient with lung ultrasonography in cardiac anaesthesiologist after training lung ultrasonography
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy
Number analyzed (Participants) | 97 | 98
Participants | 89 | 83

ADVERSE EVENTS:
Time Frame: Total intraoperative period, an average of 1 hour
Description: Desaturation
Arm/Group | Ultrasonography | Fiberoptic Bronchoscopy
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/98
Other Adverse Events (participants affected / at risk) | 33/97 | 29/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasonography (N=97) | Fiberoptic Bronchoscopy (N=98)
Hypotension (Cardiac disorders) | 33 (33) | 29 (29) — Blood pressure less than 20% of baseline
Desaturation (Cardiac disorders) | 16 (16) | 11 (11) — oxygen saturation less than 90% at any time

LIMITATIONS AND CAVEATS:
Ultrasonographer needs to be completely blind due to clinical visualization of chest rising after intubation before and during perform ultrasonography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-02-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT03314519/SAP_002.pdf
  • Study Protocol (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03314519/Prot_004.pdf